CLINICAL TRIAL: NCT03463174
Title: A Randomized Controlled Clinical Trial Alongside a Cost-effectiveness Analysis of the Mandibular Conventional Complete Denture Versus Single-implant Mandibular Overdenture
Brief Title: Cost-effectiveness of the Single-implant Mandibular Overdenture Versus Mandibular Conventional Denture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Goias (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Cláudio Rodrigues Leles, Associate professor, Universidade Federal de Goias
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UFG_020_12
Record Dates: First submitted 2018-03-05; First posted 2018-03-13 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Mouth, Edentulous; Complete Edentulism
Keywords: overdenture; edentulism; dental implant; cost-effectiveness; economic analysis; effectiveness
MeSH Terms: conditions — Mouth, Edentulous | interventions — Dental Implants; Denture, Complete

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single-implant mandibular overdenture (Experimental): Participants allocated to this group will have a dental implant placed in the mandibular midline followed by the immediately insertion of a ball attachment and the incorporation of a retention matrix to the mandibular denture.
  Interventions: Procedure: Mandibular overdenture
- Mandibular complete denture (Active Comparator): Participants allocated to this group will not receive any additional treatment besides the new set of conventional complete dentures. When needed, retreatment or any adjustment/repair in the dentures will be performed accordingly. Participants will receive regular maintenance for their dentures, including adjustments for the elimination of sore areas, denture relining and repair of fractures, when needed, until the end of the follow-up period.
  Interventions: Other: Mandibular complete denture

INTERVENTIONS:
Procedure: Mandibular overdenture — Placement of an implant in the mandibular midline.
  Other Names: Dental Implant (Straumann StandardPlus SLActive® RN implant)
  Arms: Single-implant mandibular overdenture
Other: Mandibular complete denture — No intervention.
  Other Names: Complete denture
  Arms: Mandibular complete denture

SUMMARY:
This is a randomized clinical trial designed to assess the 1-year effectiveness of two treatment modalities for the mandibular edentulists: conventional complete dentures and single-implant mandibular overdenture.

DETAILED DESCRIPTION:
This randomized clinical trial alongside a cost-effectiveness analysis will include edentulous individuals who meet eligibility criteria. New maxillary and mandibular dentures will be fabricated for all participants following a standardized protocol. Then, participants will be randomized into one of the treatment groups: conventional complete denture group or single-implant mandibular overdenture group. Each participant allocated to the overdenture group will then receive an implant (Titamax TI cortical - Neodent, Brazil) in the mandibular midline followed by the immediate connection of an O-Ring/ball attachment with intra-oral incorporation of the retention system in the mandibular denture. Direct costs related to therapies in both groups will be identified, measured and valuated for one year after treatment and patient-reported outcomes will be assessed. Incremental cost-effectiveness ratios will be estimated and graphically presented on cost-effectiveness planes. A Markov decision tree will be constructed to set out the consequences of the competing alternatives. Sensitivity analysis on the most important assumptions will be performed in order to assess the robustness of the model.

ELIGIBILITY:
Inclusion Criteria:

* To present favorable general health and the need to be rehabilitated with a new set of complete dentures
* To agree to be randomly assigned to one of the two study groups
* To be able to comprehend and answer the data collection instruments.

Exclusion Criteria:

* Presence of general health conditions that may contraindicate implant surgery (such as uncontrolled type II diabetes mellitus or uncontrolled cardiovascular conditions)
* Insufficient height and volume in the midline region to receive an implant of at least 3.75mm x 9.0mm
* Presence of evident signs of cognitive impairment and/or oral conditions requiring additional treatments, such as oral lesions and temporomandibular disorders
* Inability to attend to the scheduled appointments and follow-up visits

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-03-10 (Actual); Primary Completion 2017-09-20 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Oral health-related quality of life (OHRQoL) | From baseline to 12 months after the intervention
  The cross-culturally adapted Brazilian version of the Oral Health Impact Profile for edentulous subjects (OHIP-EDENT) will be used. It contains 19 items divided in four different subscale domains: (I) masticatory discomfort and disability (four items), (II) psychological discomfort and disability (five items), (III) social disability (five items), and (IV) oral pain and discomfort (five items). The items are answerable by a 3-point Likert scale and responses will be summed to result an overall score. Higher scores represent worse OHRQoL.

SECONDARY OUTCOMES:
Satisfaction with the dentures | From baseline to 12 months after the intervention
  Participants will report how satisfied they are on a 0-100 scale by choosing a multiple of 10. Zero will be considered the least satisfied possible and "100" the most satisfied possible.

OTHER OUTCOMES:
Costs | From denture's fabrication to 12 months after the intervention
  All the direct dental costs related to the clinical and laboratory phases of both treatment groups will be listed, measured and valued.

CONTACTS AND LOCATIONS:
Overall Officials: Claudio R Leles, DDS, PhD, Study Director — Universidade Federal de Goias
Locations (1):
- School of Dentistry, Federal University of Goias, Goiânia, Goiás, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Nogueira TE, Aguiar FMO, Esfandiari S, Leles CR. Effectiveness of immediately loaded single-implant mandibular overdentures versus mandibular complete dentures: A 1-year follow-up of a randomized clinical trial. J Dent. 2018 Oct;77:43-50. doi: 10.1016/j.jdent.2018.07.006. Epub 2018 Jul 10. PMID 30006117